CLINICAL TRIAL: NCT01632670
Title: FEAT: Functional Change in Endothelium After Cardiac cAtheterization, With and Without Music Therapy
Brief Title: Functional Change in Endothelium After Cardiac cAtheterization, With and Without Music Therapy
Acronym: FEAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emmanouil Brilakis (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Emmanouil Brilakis, Director, Cardiac Catheterization Laboratories, North Texas Veterans Healthcare System
Organization: North Texas Veterans Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-027
Record Dates: First submitted 2012-06-17; First posted 2012-07-03 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease; Endothelial Dysfunction
Keywords: music; cardiac catheterization; endothelial function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music therapy (Experimental): The music played will be by MusiCure, by Niels Eje (slow, relaxing music designed for therapeutic use), and will be played from an audio pillow beneath the patient's head.
  Interventions: Other: Music therapy
- No music therapy (No Intervention)

INTERVENTIONS:
Other: Music therapy — The music played will be by MusiCure, by Niels Eje (slow, relaxing music designed for therapeutic use), and will be played from an audio pillow beneath the patient's head.
  Arms: Music therapy

SUMMARY:
The purpose of this study is to determine the effect of music therapy before, during, and after cardiac catheterization is associated on (a) change in reactive hyperemia index measured before and after catheterization using peripheral arterial tonometry and (b) patient stress and discomfort measured by a questionnaire, as compared to the standard of care (no music during cardiac catheterization).

The hypothesis of the study is that music therapy during cardiac catheterization will be associated with more favorable change in reactive hyperemia and higher patient satisfaction compared to no music playback.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Referred for clinically-indicated cardiac catheterization

Exclusion Criteria:

1. Refusal or inability to provide signed informed consent
2. Significant hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
change in reactive hyperemia index measured by peripheral arterial tonometry | PAT will be performed within 2 hours before cardiac catheterizaiton and repeated within 2 hours after the end of cardiac catheterization

SECONDARY OUTCOMES:
Stress and anxiety questionnaire | questionnaire will be completed within 2 hours after the end of cardiac catheterization
  a stess and anxiety questionnaire will be completed within 2 hours after cardiac catheterization is completed

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Principal Investigator — North Texas Veterans Healthcare System
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States